CLINICAL TRIAL: NCT06180954
Title: A Phase I, Open-label, Two-part Study of the Absorption, Metabolism, Excretion, and the Absolute Bioavailability of [14C]-LOXO-305 in Healthy Male Subjects
Brief Title: A Study of Carbon-14-Labelled [14C] LOXO-305 (Pirtobrutinib) in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Loxo Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: LOXO-BTK-20007; J2N-OX-JZNB (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-12-13; First posted 2023-12-26 (Actual); Results first posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-11

CONDITIONS: Healthy
MeSH Terms: interventions — pirtobrutinib

STUDY DESIGN:
Intervention Model Description: This is a 2-part study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: [14C]-LOXO-305 Oral Solution (Experimental): Participants received a single dose of 200 milligram (mg) LOXO-305 radiolabelled with carbon-14, i.e., [14C]-LOXO-305 (approximately 200 microcurie radioactivity) administered as an oral solution.
  Interventions: Drug: [14C]-LOXO-305
- Part 2: LOXO-305 Oral Tablet + [14C]-LOXO-305 IV Solution (Experimental): Participants received:
  a single dose of 200 mg LOXO-305 administered as 2×100 mg oral tablets followed 2 hours later by a single dose of less than 100 microgram (μg) of [14C]-LOXO-305 (approximately 1 microcurie radioactivity) administered as an intravenous (IV) push over approximately 2 minutes.
  Interventions: Drug: LOXO-305; Drug: [14C]-LOXO-305

INTERVENTIONS:
Drug: [14C]-LOXO-305 — Administered orally
  Other Names: LY3527727
  Arms: Part 1: [14C]-LOXO-305 Oral Solution
Drug: LOXO-305 — Administered orally
  Other Names: Pirtobrutinib; LY3527727
  Arms: Part 2: LOXO-305 Oral Tablet + [14C]-LOXO-305 IV Solution
Drug: [14C]-LOXO-305 — Administered IV
  Other Names: LY3527727
  Arms: Part 2: LOXO-305 Oral Tablet + [14C]-LOXO-305 IV Solution

SUMMARY:
The main purpose of this study is to evaluate the absorption, metabolism, and excretion (AME) profiles of pirtobrutinib (LOXO-305), to identify and characterize metabolites of pirtobrutinib (LOXO-305), and to assess the safety and tolerability of [14C] LOXO-305 in Part 1. To determine the absolute bioavailability of pirtobrutinib (LOXO-305), to evaluate the plasma concentration of total radioactivity, to evaluate the urinary excretion of [14C] LOXO-305 and total radioactivity, to evaluate the fecal excretion of [14C] LOXO-305 and total radioactivity, and to assess the safety and tolerability of pirtobrutinib (LOXO-305), and [14C] LOXO-305 in Part 2. Blood tests will be performed to check how much pirtobrutinib (LOXO-305) and [14C] LOXO-305 gets into the bloodstream and how long it takes the body to eliminate it.

The study will last up to approximately 60 days for Part 1 and approximately 47 days for Part 2.

ELIGIBILITY:
Inclusion Criteria:

* Must have Body mass index (BMI) within the range of 18.5 to 32.0 kilograms per square meter (kg/m²), inclusive
* Male participants in good health, determined by no clinically significant findings from medical history, 12-lead Electrocardiogram (ECG), vital sign measurements, or clinical laboratory evaluations as assessed by the investigator
* Participants who are capable of fathering a child must agree to use contraception from the time of the dose administration through 6 months after the last dose of LOXO-305 administration
* History of a minimum of 1 bowel movement per day

Exclusion Criteria:

* History or presence of any diseases or conditions of clinical significance by the Investigator (or designee) and/or Sponsor
* Positive serologic test for hepatitis B surface antigen (HBsAg), hepatitis B virus (HBV) core antibody, hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) antibody at Screening
* Positive polymerase chain reaction (PCR) test for COVID-19 at Screening or Check-in (Day -1)
* Known ongoing alcohol and/or drug abuse within 2 years prior to Screening
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee)
* Part 1 only: Participation in a radiolabeled drug study where exposures are known to the Investigator (or designee) within the previous 4 months prior to Check-in (Day -1) or participation in a radiolabeled drug study where exposures are not known to the Investigator (or designee) within the previous 6 months prior to Check-in (Day -1).
* Part 2 only: Participation in any other radiolabeled investigational study drug trial within 12 months prior to Check-in (Day -1). Any previous radiolabeled study drug must have been received more than 12 months prior to Check-in (Day -1).

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 9 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2020-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renee Ward, MD, PhD, Study Director — Loxo Oncology, Inc.
Locations (1):
- Covance Clinical Research Unit, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 2: LOXO-305 Oral Tablet + [14C]-LOXO-305 IV Solution: Participants received:
  * a single dose of 200 mg LOXO-305 administered as 2×100 mg oral tablets
  * followed 2 hours later by a single dose of less than 100 microgram (μg) of [14C]-LOXO-305 (approximately 1 microcurie radioactivity) administered as an intravenous (IV) push over approximately 2 minutes.
Period: Overall Study
Arm/Group | Part 1: [14C]-LOXO-305 Oral Solution | Part 2: LOXO-305 Oral Tablet + [14C]-LOXO-305 IV Solution
Started | 4 | 5
Received at Least One Dose of Study Drug. | 4 | 5
Completed | 4 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Part 1: [14C]-LOXO-305 Oral Solution: Participants received a single dose of 200 mg LOXO-305 radiolabelled with carbon-14, i.e., [14C]-LOXO-305 (approximately 200 microcurie radioactivity) administered as an oral solution.
- Part 2: LOXO-305 Oral Tablet + [14C]-LOXO-305 IV Solution: Participants received:
  * a single dose of 200 mg LOXO-305 administered as 2×100 mg oral tablets
  * followed 2 hours later by a single dose of less than 100 μg of [14C]-LOXO-305 (approximately 1 microcurie radioactivity) administered as an IV push over approximately 2 minutes.
- Total: Total of all reporting groups
Arm/Group | Part 1: [14C]-LOXO-305 Oral Solution | Part 2: LOXO-305 Oral Tablet + [14C]-LOXO-305 IV Solution | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.5 (3.42) | 24 (5.15) | 30.9 (9.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 4 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 4 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 3 | 4 | 7
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Pharmacokinetics (PK): Area Under the Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC0-inf) of LOXO-305 in Plasma Following a Single Oral Dose of [14C]-LOXO-305
Description: AUC0-inf of LOXO-305 in plasma.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, 288, 312, 336, 360 hours post-dose
Population: All part 1 participants who received [14C]-LOXO-305 and had at least 1 quantifiable PK concentration, and for whom at least 1 PK parameter was computed. Participants were excluded from the analysis if they had an AE of vomiting that occurred at or before 2 times the median time to maximum observed plasma concentration (Tmax).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanogram per milliliter (h*ng/mL)
Arm/Group | Part 1: [14C]-LOXO-305 Oral Solution
Number analyzed (Participants) | 4
hours*nanogram per milliliter (h*ng/mL) | 75300 (14.8)

2. Primary Outcome: Part 1: PK: Area Under the Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC0-inf) of Total Radioactivity in Plasma and Whole Blood Following a Single Oral Dose of [14C]-LOXO-305
Description: AUC0-inf of total radioactivity in plasma and whole blood.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanogram equivalent per gram
Arm/Group | Part 1: [14C]-LOXO-305 Oral Solution
Number analyzed (Participants) | 4
hours*nanogram equivalent per gram
  Plasma | 111000 (15.8)
  Whole Blood | 71200 (12.6)

3. Primary Outcome: Part 1: PK: Area Under the Concentration-time Curve From Hour 0 to the Last Measurable Concentration (AUC0-t) of LOXO-305 in Plasma Following a Single Oral Dose of [14C]-LOXO-305
Description: AUC0-t of LOXO-305 in plasma.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanogram per milliliter (h*ng/mL)
Arm/Group | Part 1: [14C]-LOXO-305 Oral Solution
Number analyzed (Participants) | 4
hours*nanogram per milliliter (h*ng/mL) | 74500 (14.9)

4. Primary Outcome: Part 1: PK: Area Under the Concentration-time Curve From Hour 0 to the Last Measurable Concentration (AUC0-t) of Total Radioactivity in Plasma and Whole Blood Following a Single Oral Dose of [14C]-LOXO-305
Description: AUC0-t of total radioactivity in plasma and whole blood.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanogram equivalent per gram
Arm/Group | Part 1: [14C]-LOXO-305 Oral Solution
Number analyzed (Participants) | 4
hours*nanogram equivalent per gram
  Plasma | 109000 (16.1)
  Whole Blood | 68900 (13)

5. Primary Outcome: Part 1: PK: Maximum Observed Plasma Concentration (Cmax) of LOXO-305 in Plasma Following a Single Oral Dose of [14C]-LOXO-305
Description: Cmax of LOXO-305 in plasma.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Part 1: [14C]-LOXO-305 Oral Solution
Number analyzed (Participants) | 4
nanograms per milliliter (ng/mL) | 3530 (8.8)

6. Primary Outcome: Part 1: PK: Maximum Observed Plasma Concentration (Cmax) of Total Radioactivity in Plasma and Whole Blood Following a Single Oral Dose of [14C]-LOXO-305
Description: Cmax of total radioactivity in plasma and whole blood.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram equivalent per gram
Arm/Group | Part 1: [14C]-LOXO-305 Oral Solution
Number analyzed (Participants) | 4
nanogram equivalent per gram
  Plasma | 4280 (7.7)
  Whole Blood | 3020 (7.7)

7. Primary Outcome: Part 1: PK: Time to Maximum Observed Concentration (Tmax) of LOXO-305 in Plasma Following a Single Oral Dose of [14C]-LOXO-305
Description: Tmax of LOXO-305 in plasma.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Part 1: [14C]-LOXO-305 Oral Solution
Number analyzed (Participants) | 4
hours | 1.80 [1.5 to 3]

8. Primary Outcome: Part 1: PK: Time to Maximum Observed Concentration (Tmax) of Total Radioactivity in Plasma and Whole Blood Following a Single Oral Dose of [14C]-LOXO-305
Description: Tmax of total radioactivity in plasma and whole blood.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Part 1: [14C]-LOXO-305 Oral Solution
Number analyzed (Participants) | 4
hours
  Plasma | 1.80 [1.50 to 4]
  Whole Blood | 1.80 [1.50 to 3]

9. Primary Outcome: Part 1: PK: Apparent Terminal Elimination Half-life (t1/2) of LOXO-305 in Plasma Following a Single Oral Dose of [14C]-LOXO-305
Description: t1/2 of LOXO-305 in plasma.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part 1: [14C]-LOXO-305 Oral Solution
Number analyzed (Participants) | 4
hours | 17.8 (2.26)

10. Primary Outcome: Part 1: PK: Apparent Terminal Elimination Half-life (t1/2) of Total Radioactivity in Plasma and Whole Blood Following a Single Oral Dose of [14C]-LOXO-305
Description: t1/2 of total radioactivity in plasma and whole blood.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part 1: [14C]-LOXO-305 Oral Solution
Number analyzed (Participants) | 4
hours
  Plasma | 25.3 (4.76)
  Whole Blood | 21.7 (3.08)

11. Primary Outcome: Part 1: PK: Apparent Systemic Clearance (CL/F) of LOXO-305 in Plasma Following a Single Oral Dose of [14C]-LOXO-305
Description: CL/F of LOXO-305 in plasma.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/h)
Arm/Group | Part 1: [14C]-LOXO-305 Oral Solution
Number analyzed (Participants) | 4
liter per hour (L/h) | 2.69 (15.8)

12. Primary Outcome: Part 1: PK: Apparent Volume of Distribution (Vz/F) of LOXO-305 in Plasma Following a Single Oral Dose of [14C]-LOXO-305
Description: Vz/F of LOXO-305 in plasma.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter (L)
Arm/Group | Part 1: [14C]-LOXO-305 Oral Solution
Number analyzed (Participants) | 4
liter (L) | 68.8 (21)

13. Primary Outcome: Part 1: PK: Ratio of AUC0-inf of Plasma LOXO-305 to AUC0-inf of Plasma Total Radioactivity
Description: AUC0-inf of plasma LOXO-305 relative to AUC0-inf of plasma total radioactivity, expressed in ratio.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Part 1: [14C]-LOXO-305 Oral Solution
Number analyzed (Participants) | 4
ratio | 0.680 (1.2)

14. Primary Outcome: Part 1: PK: Ratio of AUC0-inf of Whole Blood Total Radioactivity to AUC0-inf of Plasma Total Radioactivity
Description: AUC0-inf of whole blood total radioactivity relative to AUC0-inf of plasma total radioactivity, expressed in ratio.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Part 1: [14C]-LOXO-305 Oral Solution
Number analyzed (Participants) | 4
ratio | 0.642 (3.4)

15. Primary Outcome: Part 1: PK: Cumulative Amount of Total Radioactivity Excreted in Urine
Description: The urine sampling time points from pre-dose through 360 hours post-dose were used to assess this outcome.
Time Frame: Pre-dose, 0 (time of dose), 6, 12, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, 288, 312, 336, 360 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligram equivalent (mg eq)
Arm/Group | Part 1: [14C]-LOXO-305 Oral Solution
Number analyzed (Participants) | 4
milligram equivalent (mg eq) | 116 (4.05)

16. Primary Outcome: Part 1: PK: Cumulative Amount of Total Radioactivity Excreted in Feces
Description: The feces sampling time points from the 0 hour (i.e. time of dose) through 360 hours post-dose were used to assess this outcome.
Time Frame: 0 (time of dose), 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, 288, 312, 336, 360 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligram equivalent (mg eq)
Arm/Group | Part 1: [14C]-LOXO-305 Oral Solution
Number analyzed (Participants) | 4
milligram equivalent (mg eq) | 75.5 (5.29)

17. Primary Outcome: Part 1: PK: Mean Cumulative Percentage of Total Radioactivity Excreted in Feces
Description: as for outcome 16
Time Frame: 0 (time of dose), 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, 288, 312, 336, 360 hours post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of total radioactivity
Arm/Group | Part 1: [14C]-LOXO-305 Oral Solution
Number analyzed (Participants) | 4
percentage of total radioactivity | 37.3 (2.31)

18. Primary Outcome: Part 1: PK: Mean Cumulative Percentage of Total Radioactivity Excreted in Urine
Description: The urine sampling time points from pre-dose through 360 hours post-dose were used to assess this outcome.
Time Frame: as for outcome 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of total radioactivity
Arm/Group | Part 1: [14C]-LOXO-305 Oral Solution
Number analyzed (Participants) | 4
percentage of total radioactivity | 57 (2.16)

19. Primary Outcome: Part 1: PK: Metabolic Profile of LOXO-305 in Plasma Following a Single Oral Dose of [14C]-LOXO-305
Description: The metabolic profile of LOXO-305 following a single oral dose of [14C]-LOXO-305 was done to assess the presence of LOXO-305 and various metabolites (M1 to M4, M11, M12, M15 to M22) in plasma using high-performance liquid chromatography with radiochemical detection. Metabolites are identified by comparison with known standards (when available) and/or by liquid chromatography/tandem mass spectrometry analysis. The presence of any metabolite in a given matrix is indicated as '1' and absence from that matrix is indicated as '0'.
Time Frame: 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264 h post-dose
Population: as for outcome 1
Measure: Number; unit: sample positive
Arm/Group | Part 1: [14C]-LOXO-305 Oral Solution
Number analyzed (Participants) | 4
sample positive
  Loxo-305 | 1
  M1 | 1
  M2 | 1
  M3 | 0
  M4 | 1
  M11 | 0
  M12 | 0
  M15 | 0
  M16 | 0
  M17 | 0
  M18 | 0
  M19 | 0
  M20 | 0
  M21 | 0
  M22 | 0

20. Primary Outcome: Part 1: PK: Metabolic Profile of LOXO-305 in Urine Following a Single Oral Dose of [14C]-LOXO-305
Description: The metabolic profile of LOXO-305 following a single oral dose of [14C]-LOXO-305 was done to assess the presence of LOXO-305 and various metabolites (M1 to M4, M11, M12, M15 to M22) in urine using high-performance liquid chromatography with radiochemical detection. Metabolites are identified by comparison with known standards (when available) and/or by liquid chromatography/tandem mass spectrometry analysis. The presence of any metabolite in a given matrix is indicated as '1' and absence from that matrix is indicated as '0'.
Time Frame: as for outcome 15
Population: as for outcome 1
Measure: Number; unit: sample positive
Arm/Group | Part 1: [14C]-LOXO-305 Oral Solution
Number analyzed (Participants) | 4
sample positive
  Loxo-305 | 1
  M1 | 0
  M2 | 1
  M3 | 1
  M4 | 1
  M11 | 0
  M12 | 1
  M15 | 1
  M16 | 1
  M17 | 1
  M18 | 1
  M19 | 1
  M20 | 0
  M21 | 0
  M22 | 0

21. Primary Outcome: Part 1: PK: Metabolic Profile of LOXO-305 in Feces Following a Single Oral Dose of [14C]-LOXO-305
Description: The metabolic profile of LOXO-305 following a single oral dose of [14C]-LOXO-305 was done to assess the presence of LOXO-305 and various metabolites (M1 to M4, M11, M12, M15 to M22) in feces using high-performance liquid chromatography with radiochemical detection. Metabolites are identified by comparison with known standards (when available) and/or by liquid chromatography/tandem mass spectrometry analysis. The presence of any metabolite in a given matrix is indicated as '1' and absence from that matrix is indicated as '0'.
Time Frame: 0 (time of dose), 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, 288, 312, 336, 360 hours post-dose
Population: as for outcome 1
Measure: Number; unit: sample positive
Arm/Group | Part 1: [14C]-LOXO-305 Oral Solution
Number analyzed (Participants) | 4
sample positive
  Loxo-305 | 1
  M1 | 0
  M2 | 0
  M3 | 0
  M4 | 0
  M11 | 1
  M12 | 0
  M15 | 0
  M16 | 1
  M17 | 0
  M18 | 0
  M19 | 0
  M20 | 1
  M21 | 1
  M22 | 1

22. Primary Outcome: Part 2: PK: Area Under the Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC0-inf) of LOXO-305 in Plasma
Description: AUC0-inf of LOXO-305 in plasma. The sampling time points from pre-oral dose through 192 hours post-IV dose were used to assess this outcome.
Time Frame: Pre-oral dose, 0.5, 1, 2 hours post oral dose, 0.03, 0.17, 0.33, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, 168, 192 hours post IV dose.
Population: All part 2 participants who received LOXO-305 and had at least 1 quantifiable PK concentration, and for whom at least 1 PK parameter was computed. Participants were excluded from the analysis if they had an AE of vomiting that occurred at or before 2 times the median time to maximum observed plasma concentration (Tmax).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanogram per milliliter (h*ng/mL)
Arm/Group | Part 2: LOXO-305 Oral Tablet + [14C]-LOXO-305 IV Solution
Number analyzed (Participants) | 5
hours*nanogram per milliliter (h*ng/mL) | 105000 (28.1)

23. Primary Outcome: Part 2: PK: Area Under the Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC0-inf) of [14C]-LOXO-305 in Plasma
Description: AUC0-inf of [14C]-LOXO-305 in plasma. The sampling time points from pre-IV dose through 192 hours post-IV dose were used to assess this outcome.
Time Frame: Pre-IV dose, 0.03, 0.17, 0.33, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 96, 120, 144, 168, 192 hours post IV dose.
Population: All part 2 participants who received [14C]-LOXO-305 and had at least 1 quantifiable PK concentration, and for whom at least 1 PK parameter was computed. Participants were excluded from the analysis if they had an AE of vomiting that occurred at or before 2 times the median time to maximum observed plasma concentration (Tmax).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*picogram per milliliter
Arm/Group | Part 2: LOXO-305 Oral Tablet + [14C]-LOXO-305 IV Solution
Number analyzed (Participants) | 5
hours*picogram per milliliter | 13700 (29)

24. Primary Outcome: Part 2: PK: Area Under the Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC0-inf) of Total Radioactivity in Plasma
Description: AUC0-inf of total radioactivity in plasma. The sampling time points from pre-IV dose through 192 hours post-IV dose were used to assess this outcome.
Time Frame: as for outcome 23
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*picogram equivalent per milliliter
Arm/Group | Part 2: LOXO-305 Oral Tablet + [14C]-LOXO-305 IV Solution
Number analyzed (Participants) | 5
hours*picogram equivalent per milliliter | 18300 (25.2)

25. Primary Outcome: Part 2: PK: Area Under the Concentration-time Curve From Hour 0 to the Last Measurable Concentration (AUC0-t) of LOXO-305 in Plasma
Description: AUC0-t of LOXO-305 in plasma. The sampling time points from pre-oral dose through 192 hours post-IV dose were used to assess this outcome.
Time Frame: as for outcome 22
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanogram per milliliter (h*ng/mL)
Arm/Group | Part 2: LOXO-305 Oral Tablet + [14C]-LOXO-305 IV Solution
Number analyzed (Participants) | 5
hours*nanogram per milliliter (h*ng/mL) | 104000 (28.7)

26. Primary Outcome: Part 2: PK: Area Under the Concentration-time Curve From Hour 0 to the Last Measurable Concentration (AUC0-t) of [14C]-LOXO-305 in Plasma
Description: AUC0-t of [14C]-LOXO-305 in plasma. The sampling time points from pre-IV dose through 192 hours post-IV dose were used to assess this outcome.
Time Frame: as for outcome 23
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*picogram per milliliter
Arm/Group | Part 2: LOXO-305 Oral Tablet + [14C]-LOXO-305 IV Solution
Number analyzed (Participants) | 5
hours*picogram per milliliter | 13700 (29.2)

27. Primary Outcome: Part 2: PK: Area Under the Concentration-time Curve From Hour 0 to the Last Measurable Concentration (AUC0-t) of Total Radioactivity in Plasma
Description: AUC0-t of Total Radioactivity in Plasma. The sampling time points from pre-IV dose through 192 hours post-IV dose were used to assess this outcome.
Time Frame: as for outcome 23
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*picogram equivalent per milliliter
Arm/Group | Part 2: LOXO-305 Oral Tablet + [14C]-LOXO-305 IV Solution
Number analyzed (Participants) | 5
hours*picogram equivalent per milliliter | 18000 (25.8)

28. Primary Outcome: Part 2: PK: Maximum Observed Plasma Concentration (Cmax) of LOXO-305 in Plasma
Description: Cmax of LOXO-305 in plasma. The sampling time points from pre-oral dose through 192 hours post-IV dose were used to assess this outcome.
Time Frame: as for outcome 22
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Part 2: LOXO-305 Oral Tablet + [14C]-LOXO-305 IV Solution
Number analyzed (Participants) | 5
nanograms per milliliter (ng/mL) | 4490 (19.2)

29. Primary Outcome: Part 2: PK: Maximum Observed Plasma Concentration (Cmax) of [14C]-LOXO-305 in Plasma
Description: Cmax of [14C]-LOXO-305 in plasma. The sampling time points from pre-IV dose through 192 hours post-IV dose were used to assess this outcome.
Time Frame: as for outcome 23
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram per milliliter (pg/mL)
Arm/Group | Part 2: LOXO-305 Oral Tablet + [14C]-LOXO-305 IV Solution
Number analyzed (Participants) | 5
picogram per milliliter (pg/mL) | 994 (31.6)

30. Primary Outcome: Part 2: PK: Maximum Observed Plasma Concentration (Cmax) of Total Radioactivity in Plasma
Description: Cmax of Total Radioactivity in Plasma. The sampling time points from pre-IV dose through 192 hours post-IV dose were used to assess this outcome.
Time Frame: as for outcome 23
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram equivalent per milliliter
Arm/Group | Part 2: LOXO-305 Oral Tablet + [14C]-LOXO-305 IV Solution
Number analyzed (Participants) | 5
picogram equivalent per milliliter | 1110 (53.1)

31. Primary Outcome: Part 2: PK: Time to Maximum Observed Concentration (Tmax) of LOXO-305 in Plasma
Description: Tmax of LOXO-305 in plasma. The sampling time points from pre-oral dose through 192 hours post-IV dose were used to assess this outcome.
Time Frame: as for outcome 22
Population: as for outcome 22
Measure: Median (Full Range); unit: hours
Arm/Group | Part 2: LOXO-305 Oral Tablet + [14C]-LOXO-305 IV Solution
Number analyzed (Participants) | 5
hours | 5.00 [2.03 to 5]

32. Primary Outcome: Part 2: PK: Time to Maximum Observed Concentration (Tmax) of [14C]-LOXO-305 in Plasma
Description: Tmax of [14C]-LOXO-305 in plasma. The sampling time points from pre-IV dose through 192 hours post-IV dose were used to assess this outcome.
Time Frame: as for outcome 23
Population: as for outcome 23
Measure: Median (Full Range); unit: hours
Arm/Group | Part 2: LOXO-305 Oral Tablet + [14C]-LOXO-305 IV Solution
Number analyzed (Participants) | 5
hours | 0.167 [0.0333 to 12]

33. Primary Outcome: Part 2: PK: Time to Maximum Observed Concentration (Tmax) of Total Radioactivity in Plasma
Description: Tmax of Total Radioactivity in plasma. The sampling time points from pre-IV dose through 192 hours post-IV dose were used to assess this outcome.
Time Frame: as for outcome 23
Population: as for outcome 23
Measure: Median (Full Range); unit: hours
Arm/Group | Part 2: LOXO-305 Oral Tablet + [14C]-LOXO-305 IV Solution
Number analyzed (Participants) | 5
hours | 0.167 [0.0333 to 0.167]

34. Primary Outcome: Part 2: PK: Apparent Terminal Elimination Half-life (t1/2) of LOXO-305 in Plasma
Description: t1/2 of LOXO-305 in plasma. The sampling time points from pre-oral dose through 192 hours post-IV dose were used to assess this outcome.
Time Frame: as for outcome 22
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part 2: LOXO-305 Oral Tablet + [14C]-LOXO-305 IV Solution
Number analyzed (Participants) | 5
hours | 18.7 (1.68)

35. Primary Outcome: Part 2: PK: Apparent Terminal Elimination Half-life (t1/2) of [14C]-LOXO-305 in Plasma
Description: t1/2 of [14C]-LOXO-305 in plasma. The sampling time points from pre-IV dose through 192 hours post-IV dose were used to assess this outcome.
Time Frame: as for outcome 23
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part 2: LOXO-305 Oral Tablet + [14C]-LOXO-305 IV Solution
Number analyzed (Participants) | 5
hours | 17.6 (1.24)

36. Primary Outcome: Part 2: PK: Apparent Terminal Elimination Half-life (t1/2) of Total Radioactivity in Plasma
Description: t1/2 of Total Radioactivity in plasma. The sampling time points from pre-IV dose through 192 hours post-IV dose were used to assess this outcome.
Time Frame: as for outcome 23
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part 2: LOXO-305 Oral Tablet + [14C]-LOXO-305 IV Solution
Number analyzed (Participants) | 5
hours | 37.4 (9.72)

37. Primary Outcome: Part 2: PK: Apparent Systemic Clearance (CL/F) of LOXO-305 in Plasma
Description: CL/F of LOXO-305 in plasma. The sampling time points from pre-oral dose through 192 hours post-IV dose were used to assess this outcome.
Time Frame: as for outcome 22
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/h)
Arm/Group | Part 2: LOXO-305 Oral Tablet + [14C]-LOXO-305 IV Solution
Number analyzed (Participants) | 5
liter per hour (L/h) | 1.90 (28.1)

38. Primary Outcome: Part 2: PK: Apparent Volume of Distribution During the Terminal Phase (Vz/F) of LOXO-305 in Plasma
Description: Vz/F of LOXO-305 in plasma. The sampling time points from pre-oral dose through 192 hours post-IV dose were used to assess this outcome.
Time Frame: as for outcome 22
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter (L)
Arm/Group | Part 2: LOXO-305 Oral Tablet + [14C]-LOXO-305 IV Solution
Number analyzed (Participants) | 5
liter (L) | 51.0 (23.6)

39. Primary Outcome: Part 2: PK: Absolute Bioavailability of LOXO-305 in Plasma
Description: The absolute bioavailability expressed in ratio was calculated using the formula= AUC0-inf (oral) x Dose (IV) divided by AUC0-inf (IV) x Dose (oral) . The sampling time points from pre-oral dose through 192 hours post-IV dose were used to assess this outcome.
Time Frame: as for outcome 22
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Part 2: LOXO-305 Oral Tablet + [14C]-LOXO-305 IV Solution
Number analyzed (Participants) | 5
ratio | 0.855 (7.2)

40. Primary Outcome: Part 2: PK: Total Clearance (CL) of [14C]-LOXO-305 in Plasma
Description: CL of [14C]-LOXO-305 in plasma. The sampling time points from pre-IV dose through 192 hours post-IV dose were used to assess this outcome.
Time Frame: as for outcome 23
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/h)
Arm/Group | Part 2: LOXO-305 Oral Tablet + [14C]-LOXO-305 IV Solution
Number analyzed (Participants) | 5
liter per hour (L/h) | 1.63 (29.7)

41. Primary Outcome: Part 2: PK: Volume of Distribution (Vz) of [14C]-LOXO-305 in Plasma
Description: Vz of [14C]-LOXO-305 in plasma. The sampling time points from pre-IV dose through 192 hours post-IV dose were used to assess this outcome.
Time Frame: as for outcome 23
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter (L)
Arm/Group | Part 2: LOXO-305 Oral Tablet + [14C]-LOXO-305 IV Solution
Number analyzed (Participants) | 5
liter (L) | 41.2 (29)

42. Primary Outcome: Part 2: PK: Volume of Distribution at Steady State (Vss) of [14C]-LOXO-305 in Plasma
Description: Vss of [14C]-LOXO-305 in plasma. The sampling time points from pre-IV dose through 192 hours post-IV dose were used to assess this outcome.
Time Frame: as for outcome 23
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter (L)
Arm/Group | Part 2: LOXO-305 Oral Tablet + [14C]-LOXO-305 IV Solution
Number analyzed (Participants) | 5
liter (L) | 36.3 (24.2)

43. Primary Outcome: Part 2: PK: Renal Clearance (CLR) of [14C]-LOXO-305
Description: CLR of [14C]-LOXO-305 in urine collection. The urine sampling time points from pre-IV dose through 192 hours post-IV dose were used to assess this outcome.
Time Frame: Pre-IV dose, 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 hours post IV dose
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/h)
Arm/Group | Part 2: LOXO-305 Oral Tablet + [14C]-LOXO-305 IV Solution
Number analyzed (Participants) | 5
liter per hour (L/h) | 0.116 (36.8)

44. Primary Outcome: Part 2: PK: Cumulative Amount of [14C]-LOXO-305 Excreted in Urine
Description: The urine sampling time points from pre-oral dose through 192 hours post-IV dose were used to assess this outcome.
Time Frame: Pre-oral dose, 0 (time of oral dose), 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 hours post IV dose
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram (μg)
Arm/Group | Part 2: LOXO-305 Oral Tablet + [14C]-LOXO-305 IV Solution
Number analyzed (Participants) | 5
microgram (μg) | 1.59 (28.3)

45. Primary Outcome: Part 2: PK: Cumulative Amount of Total Radioactivity Excreted in Urine
Description: The urine sampling time points from pre-oral dose through 192 hours post-IV dose were used to assess this outcome.
Time Frame: Pre-oral dose, 0 (time of oral dose), 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 hours post IV dose
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram equivalent (μg eq)
Arm/Group | Part 2: LOXO-305 Oral Tablet + [14C]-LOXO-305 IV Solution
Number analyzed (Participants) | 5
microgram equivalent (μg eq) | 14.1 (11.4)

46. Primary Outcome: Part 2: PK: Cumulative Amount of [14C]-LOXO-305 Excreted in Feces
Description: The Feces sampling time points from the 0 hour (i.e. time of oral dose) through 192 hours post-IV dose were used to assess this outcome.
Time Frame: 0 (time of oral dose), 12, 24, 48, 72, 96, 120, 144, 168, 192 hours post IV dose
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram (μg)
Arm/Group | Part 2: LOXO-305 Oral Tablet + [14C]-LOXO-305 IV Solution
Number analyzed (Participants) | 5
microgram (μg) | 3.02 (40.5)

47. Primary Outcome: Part 2: PK: Cumulative Amount of Total Radioactivity Excreted in Feces
Description: as for outcome 46
Time Frame: 0 (time of oral dose), 12, 24, 48, 72, 96, 120, 144, 168, 192 hours post IV dose
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram equivalent (μg eq)
Arm/Group | Part 2: LOXO-305 Oral Tablet + [14C]-LOXO-305 IV Solution
Number analyzed (Participants) | 5
microgram equivalent (μg eq) | 4.97 (38.4)

48. Primary Outcome: Part 2: PK: Mean Cumulative Percentage of [14C]-LOXO-305 Excreted in Urine
Description: The urine sampling time points from pre-oral dose through 192 hours post-IV dose were used to assess this outcome.
Time Frame: Pre-oral dose, 0 (time of oral dose), 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 hours post IV dose
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of [14C]-LOXO-305
Arm/Group | Part 2: LOXO-305 Oral Tablet + [14C]-LOXO-305 IV Solution
Number analyzed (Participants) | 5
percentage of [14C]-LOXO-305 | 7.12 (28.9)

49. Primary Outcome: Part 2: PK: Mean Cumulative Percentage of Total Radioactivity Excreted in Urine
Description: The urine sampling time points from pre-oral dose through 192 hours post-IV dose were used to assess this outcome.
Time Frame: Pre-oral dose, 0 (time of oral dose), 4, 8, 12, 24, 48, 72, 96, 120, 144, 168, 192 hours post IV dose
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of total radioactivity
Arm/Group | Part 2: LOXO-305 Oral Tablet + [14C]-LOXO-305 IV Solution
Number analyzed (Participants) | 5
percentage of total radioactivity | 63.1 (11.2)

50. Primary Outcome: Part 2: PK: Mean Cumulative Percentage of [14C]-LOXO-305 Excreted in Feces
Description: as for outcome 46
Time Frame: 0 (time of oral dose), 12, 24, 48, 72, 96, 120, 144, 168, 192 hours post IV dose
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of [14C]-LOXO-305
Arm/Group | Part 2: LOXO-305 Oral Tablet + [14C]-LOXO-305 IV Solution
Number analyzed (Participants) | 5
percentage of [14C]-LOXO-305 | 13.5 (40.5)

51. Primary Outcome: Part 2: PK: Mean Cumulative Percentage of Total Radioactivity Excreted in Feces
Description: as for outcome 46
Time Frame: 0 (time of oral dose), 12, 24, 48, 72, 96, 120, 144, 168, 192 hours post IV dose
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of total radioactivity
Arm/Group | Part 2: LOXO-305 Oral Tablet + [14C]-LOXO-305 IV Solution
Number analyzed (Participants) | 5
percentage of total radioactivity | 22.3 (38.8)

ADVERSE EVENTS:
Time Frame: Part 1: Baseline up to Day 29; Part 2: Baseline up to Day 16
Description: All participants who received at least one dose of study drug. As per the planned safety analyses, AE data was reported per treatment regimen.
Groups:
- Part 2: LOXO-305 Oral Tablet + [14C]-LOXO-305 IV Solution: Participants received:
  a single dose of 200 mg LOXO-305 administered as 2×100 mg oral tablets followed 2 hours later by a single dose of less than 100 μg of [14C]-LOXO-305 (approximately 1 microcurie radioactivity) administered as an IV push over approximately 2 minutes.
Arm/Group | Part 1: [14C]-LOXO-305 Oral Solution | Part 2: LOXO-305 Oral Tablet + [14C]-LOXO-305 IV Solution
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 3/4 | 4/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: [14C]-LOXO-305 Oral Solution (N=4) | Part 2: LOXO-305 Oral Tablet + [14C]-LOXO-305 IV Solution (N=5)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Post procedural contusion (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-06-29): https://cdn.clinicaltrials.gov/large-docs/54/NCT06180954/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-13): https://cdn.clinicaltrials.gov/large-docs/54/NCT06180954/SAP_001.pdf